CLINICAL TRIAL: NCT06727708
Title: A Comparative Study of Two Biocircuit Training Programs:Tone Your Body Vs. Boost Performance on Physical Performance and Body Composition a Randomized Controlled Trial
Brief Title: Comparison of Two BioCircuit Programs: Impact on Physical Fitness and Body Composition in Adults Aged 30-65
Acronym: Biocircuit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio-RCT-2024-02
Record Dates: First submitted 2024-09-30; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-09

CONDITIONS: Muscle Strength; Body Composition; Physical Fitness
Keywords: Circle Training; Strength training; Muscle mass; Body composition; Physical fitness; BioCircuit; Resistance training; Body fat reduction; Randomized controlled trial; Handgripstrength

STUDY DESIGN:
Intervention Model Description: This trial uses a randomised parallel group design with minimisation to ensure balanced allocation based on age, gender and baseline handgrip strength. Participants will be assigned to one of two intervention groups, 'Tone Your Body' or 'Boost Performance'. Each group follows a 12-week BioCircuit training programme designed to improve physical fitness, muscle strength and body composition. Both programmes include strength and endurance exercises in a circuit format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tone Your Body Group (Experimental): Participants in the Tone Your Body group follow a 12-week BioCircuit training programme designed to improve body composition and muscle toning. The programme consists of six total-body strength exercises and two cardio exercises in a circuit format. Each exercise is performed for 45 seconds, followed by a 40-second rest between machines. The endurance exercises are performed for 3 minutes and 35 seconds each. The eccentric phase of each strength exercise is overloaded by 20% to maximise muscle development.
  Interventions: Device: Tone Your Body BioCircuit Program
- Boost Performance Group (Experimental): Participants in the Boost Performance group follow a 12-week BioCircuit training programme designed to increase strength and endurance. The programme consists of six strength exercises and two cardio exercises, also in a circuit format. Each exercise is performed for 45 seconds, with 40 seconds rest between machines, and the endurance exercises are performed for 3 minutes and 35 seconds. The strength exercises use a viscous resistance mechanism to increase strength and endurance. Participants also undergo performance tests including the jump and reach test, one minute squats and one minute push-ups.
  Interventions: Device: Boost Performance BioCircuit Program

INTERVENTIONS:
Device: Tone Your Body BioCircuit Program — Participants in the Tone Your Body group follow a 12-week BioCircuit training programme designed to improve body composition and muscle toning. The programme consists of six total-body strength exercises and two cardio exercises in a circuit format. Each exercise is performed for 45 seconds, followed by a 40-second rest between machines. The endurance exercises are performed for 3 minutes and 35 seconds each. The eccentric phase of each strength exercise is overloaded by 20% to maximise muscle development.
  Arms: Tone Your Body Group
Device: Boost Performance BioCircuit Program — Participants in the Boost Performance group follow a 12-week BioCircuit training programme designed to increase strength and endurance. The programme consists of six strength exercises and two cardio exercises, also in a circuit format. Each exercise is performed for 45 seconds, with 40 seconds rest between machines, and the endurance exercises are performed for 3 minutes and 35 seconds. The strength exercises use a viscous resistance mechanism to increase strength and endurance. Participants also undergo performance tests including the jump and reach test, one minute squats and one minute push-ups.
  Arms: Boost Performance Group

SUMMARY:
This study aims to compare the effects of two BioCircuit training programmes, 'Tone Your Body' and 'Boost Performance', on physical fitness and body composition in adults aged 30-65 years. Participants will be randomized to one of the two exercise programmes and will undergo a 12-week intervention with baseline and post-intervention measurements of fitness and body composition. The study aims to determine which programme is more effective in improving overall physical fitness, muscle mass and reducing body fat.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of two BioCircuit training programmes, 'Tone Your Body' and 'Boost Performance', on physical fitness and body composition in adults aged 30-65 years. The aim is to determine whether these programmes achieve their intended outcomes - specifically, whether Tone Your Body is effective in reducing body fat while promoting muscle toning, and whether Boost Performance improves strength and endurance. The study will assess which of the two programmes leads to greater improvements in muscle mass, body fat reduction and overall physical fitness.

The study is designed as a randomised parallel group trial using a minimisation technique to ensure that key variables such as age, gender and baseline handgrip strength are balanced between the two groups. Participants will be assigned to one of two BioCircuit programmes: "Tone Your Body" or "Boost Performance". Each programme consists of six total body strength exercises and two cardio exercises, both structured in a circuit format. Each exercise is performed for 45 seconds, followed by a 40-second rest between machines. The endurance exercises are performed for 3 minutes and 35 seconds each. The intervention will last 12 weeks, with participants training three times a week on Technogym's BioCircuit equipment, which provides personalised, automated training based on individual fitness levels.

The Tone Your Body group focuses on improving body composition through moderate-intensity whole-body resistance exercise combined with cardio training. This programme is designed to reduce body fat while promoting muscle toning, with an emphasis on overloading the eccentric phase of each repetition by 20% to maximise muscle development.

The Boost Performance group aims to improve physical performance, particularly strength and endurance. This programme involves higher intensity resistance training with a viscous resistance mechanism designed to build muscle strength, power and endurance. Participants in this group will also undergo performance tests, including the jump and reach test, one-minute squats and one-minute push-ups, to assess improvements in explosive strength and muscular endurance.

Both groups will undergo the same 10RM strength tests at baseline and post-intervention using the Smith machine for bench press and leg press to measure maximum strength. In addition, all participants, regardless of group, will undergo the same assessments at baseline and post-intervention, including measurements of body composition (using bioimpedance analysis), muscle mass, body fat percentage, and physical performance tests. Circumference measurements of the arms, legs and waist will also be taken to track changes in body composition over time. Participants will be instructed to maintain their usual dietary habits throughout the 12-week intervention period. They will be asked not to make any significant changes to their diet or to introduce any new dietary supplements, as these could influence the outcomes related to muscle strength, body composition and overall physical fitness.

The primary outcome measures will focus on changes in skeletal muscle mass, body fat percentage and overall physical fitness. Secondary outcomes will include participant satisfaction with the programme as measured by a standardised customer satisfaction questionnaire (CSAT) and changes in circumference measurements.

Participants will be healthy adults aged 30-65 years with less than six months experience of resistance training. Individuals with a history of coronary heart disease, stroke or conditions that would affect their ability to participate in exercise will be excluded from the study. Recruitment will take place through a local fitness centre and all participants will provide written informed consent before the start of the study.

This study aims to provide valuable insights into the effectiveness of BioCircuit training programmes in a real-world setting. The results will help inform future fitness interventions and provide evidence for the benefits of automated, personalised training programmes in improving body composition and physical performance in adults.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 30 and 65 years

  * Healthy individuals without significant medical conditions
  * Less than 6 months of prior strength training experience
  * Willing and able to participate in a 12-week training program
  * Capable of performing strength training exercises such as leg press and chest press
  * Able to provide written informed consent

Exclusion Criteria:

* • History of coronary heart disease

  * History of stroke
  * Need for changes in antihypertensive treatment within 3 months prior to study start
  * Arthritis
  * Pregnancy or less than three months postpartum
  * Pain and movement restrictions
  * Use of medications that affect muscle strength or performance (e.g., anabolic steroids, beta-2 agonists, glucocorticoids, statins, benzodiazepines, ACE inhibitors, angiotensin-II receptor blockers, diuretics)
  * Any medical condition preventing participation in planned endurance and strength training

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Mass | Baseline and Week 12
  Skeletal muscle mass will be measured using bioimpedance analysis (BIA) at baseline and after the 12-week intervention to evaluate changes in muscle mass.
Change in Body Fat Percentage | Baseline and Week 12
  Body fat percentage will be measured using bioimpedance analysis (BIA) at baseline and after the 12-week intervention to assess reductions in body fat.
Change in Maximal Strength (10-RM Test) | Baseline and Week 12
  Maximal strength will be measured using the 10-RM test on the Smith machine for bench press and leg press at baseline and after the 12-week intervention.
Change in Handgrip Strength | Baseline and Week 12
  Handgrip strength will be measured using a dynamometer at baseline and after the 12-week intervention.

SECONDARY OUTCOMES:
Change in Circumference Measurements (Arm, Leg, and Waist) | Baseline and Week 12
  Circumference measurements of the arms, legs, and waist will be taken at baseline and after the 12-week intervention to track changes in body composition.
Customer Satisfaction (CSAT Questionnaire) | Week 2 and Week 12
  Participant satisfaction with the training program will be assessed using the CSAT questionnaire at the end of the 12-week intervention.
Change in Jump and Reach Performance | Baseline and Week 12
  Performance will be evaluated by measuring the vertical jump height using the jump and reach test at baseline and after the 12-week intervention.
Change in Squat Performance (One-Minute Squat Test) | Baseline and Week 12
  Performance will be evaluated by counting the number of squats completed in one minute at baseline and after the 12-week intervention.
Change in Push-up Performance (One-Minute Push-up Test) | Baseline and Week 12
  Performance will be evaluated by counting the number of push-ups completed in one minute at baseline and after the 12-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Atia, Principal Investigator — University of Graz
Locations (1):
- CF Leibnitz, Leibnitz, Styria, Styria, Austria

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) used in the published results will be shared in an anonymized format. Access will be provided upon request through a secure data repository for researchers who meet the criteria for access to confidential data.
Supporting Information: Study Protocol
Time Frame: Available upon publication for one year.